CLINICAL TRIAL: NCT06465095
Title: Evaluation of Inflammasome Gene Polymorphisms in Patients With Stage III, Grade B and C Periodontitis
Brief Title: Evaluation of Inflammasome Gene Polymorphisms in Periodontitis Patients
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09-2023-1700
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-02

CONDITIONS: Periodontal Diseases; Periodontitis
Keywords: Periodontitis, gene, polymorphism
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — BaseLine dental cement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: Individuals without a clinical inflammation pattern and a history of periodontitis, with no detected clinical attachment and bone loss, BOP < 10%, probing depth ≤ 3 mm.
  Interventions: Genetic: Baseline
- Stage III Grade B Periodontitis: Individuals that have minimum of 20 teeth (except third molars), with CAL ≥ 5 mm, probing depth ≥ 6mm, and radiographically showing bone loss extending up to one-third of the root, percantage of bone lose by age is 0.25-1 will be included.
  Interventions: Genetic: Baseline
- Stage III Grade C Periodontitis: Individuals that have minimum of 20 teeth (except third molars), with CAL ≥ 5 mm, probing depth ≥ 6mm, and radiographically showing bone loss extending up to one-third of the root, percantage of bone lose by age is >1 will be included.
  Interventions: Genetic: Baseline

INTERVENTIONS:
Genetic: Baseline — Measurements and sampling

SUMMARY:
The present study aimed to evaluate the distribution of NLRP3, AIM2, and IFI16 inflammasome gene polymorphisms in individuals with Stage III Grade B and C periodontitis and periodontally healthy individuals. 80 periodontally healthy, 80 Stage III Grade B and 80 Stage III Grade C periodontitis patients will be enrolled. Blood samples will be collected from each participants and clinical parameteres will be recorded for whole mouth. DNA isolation will be performed from all samples. The SNP regions with the numbers rs4612666, rs75985579, and rs2793845 will be detected from DNA material using Real-Time PCR device genotyping kits. Data will be analyzed using statistical tests.

DETAILED DESCRIPTION:
Innate immune response is the first line of defense mechanism of the body against pathogens. One of the most important proteins involved in the innate immune response are the inflammasomes which are multimeric protein complexes composed of a sensor molecule (the PRR), typically the adapter molecule apoptosis-associated speck-like protein containing a caspase-recruitment domain (CARD), and the protease caspase-1. Different types of inflammasomes have been described. In periodontal disease, inflammasome activation is associated with the release of pro-inflammatory cytokines, which can lead to tissue destruction and periodontal damage.

Progression rate, onset age, and severity of periodontal disease are influenced by some modifiable or non-modifiable risk factors present in the host. Genetic polymorphisms are non-modifiable risk factors for periodontitis. Variations in inflammasome genes may be determinants in the development of periodontal disease by leading to diversity in inflammatory markers.

Sample size is determined based on a previous study which analyzes the effect of NLRP3 gene polymorphism on periodontitis susceptibility. For rs4612666 group, with an α value of 0.05 and a power of 80%, it is determined that there should be 80 participants in each group. Totally 240 patients are included (80 periodontally healthy, 80 Stage III Grade B periodontitis, 80 Stage III Grade C periodontitis). The whole mouth clinical periodontal examination includes measurement of probing depth (PPD), clinical attachment level (CAL), presence of bleeding on probing (BOP), gingival index (GI), and plaque index (PI) at 6 sites per tooth, except the third molars. Periodontal diagnosis of each patient has been made according to the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions. Healthy group includes individuals without a clinical inflammation pattern and a history of periodontitis, with no detected clinical attachment and bone loss, BOP < 10%, probing depth ≤ 3 mm. Stage III Grade B periodontitis patients have minimum of 20 teeth (except third molars), with CAL ≥ 5 mm, probing depth ≥ 6mm, and radiographically showing bone loss extending up to one-third of the root, percantage of bone lose by age is 0.25-1 and Stage III Grade C patients have minimum of 20 teeth (except third molars), with CAL ≥ 5 mm, probing depth ≥ 6mm, and radiographically showing bone loss extending up to one-third of the root, percantage of bone lose by age is >1.

Sample Collection and DNA Isolation and Genotyping A total of 5 mL of blood is collected from the antecubital fossa by venepuncture method from each participants and stored at -80°C until analysis day. DNA isolation has been made using genomic DNA kits. rs4612666, rs75985579, and rs2793845 SNP regions are detected from DNA material using Real-Time PCR device genotyping kits.

Statistical analysis has been performed with standard statistical software package by selecting appropriate tests.

ELIGIBILITY:
Inclusion Criteria:

* systematically healthy, non-smoker individuals
* patients between the ages of 18 and 65
* individuals with periodontally healthy, stage III grade B and C periodontitis diagnoses

Exclusion Criteria:

* having any diagnosed medical disorders such as diabetes mellitus, cardiovascular diseases, rheumatoid arthritis...
* Usage of antibiotics, non-steroidal anti-inflammatory drugs and immunosuppressive agents within the past 6 months.
* Periodontal treatment within the preceding 6 months.
* Pregnant/ lactating/ postmenopausal females.
* Current orthodontic treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sistemically healthy, non-smokers. Periorodontally healthy, stage III perodontitis B and C periodontitis patients.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-14 (Estimated); Study Completion 2025-04-14 (Estimated)

PRIMARY OUTCOMES:
NLRP3 gene polymorphism | Baseline
  SNP

SECONDARY OUTCOMES:
AIM2 gene polymorphism | Baseline
  SNP
IFI16 | Baseline
  SNP

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)